CLINICAL TRIAL: NCT05232409
Title: A Phase I Study to Determine the Safety and Recommended Phase 2 Dosing of Zeaxanthin Alone or in Combination With Pembrolizumab in Patients With Metastatic Solid Tumors
Brief Title: Determine Safety & Recommended Phase 2 Dosing of Zeaxanthin Alone or in Combination w/Pembrolizumab in Patients With Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20.0046
Record Dates: First submitted 2021-10-08; First posted 2022-02-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cancer Metastatic; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Zeaxanthins; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zeaxanthin Monotherapy (Experimental): Zeaxanthin administered orally on daily basis.
  Interventions: Biological: Zeaxanthin
- Zeaxanthin plus Pembrolizumab (Experimental): Zeaxanthin administered orally on daily basis in addition to intravenous pembrolizumab infused every 42 days at fixed dose of 400 mg.
  Interventions: Combination Product: Zeaxanthin Plus Pembrolizumab

INTERVENTIONS:
Biological: Zeaxanthin — The doses of zeaxanthin will be based on weight starting with 2 milligrams of zeaxanthin per kilogram of your body weight (mg/kg) followed by 4 mg/kg, 6 mg/kg, and finally 8 mg/kg. If a dose level is found to be unsafe, then a new group of patients will be treated at the midpoint dose between the not tolerated dose and the last tolerated dose. Zeaxanthin is supplied as 50 milligram capsules and a person's dose will be rounded to the nearest 50 milligrams.
  Arms: Zeaxanthin Monotherapy
Combination Product: Zeaxanthin Plus Pembrolizumab — The doses of zeaxanthin will be based on weight starting with 2 milligrams of zeaxanthin per kilogram of your body weight (mg/kg) followed by 4 mg/kg, 6 mg/kg, and finally 8 mg/kg. If a dose level is found to be unsafe, then a new group of patients will be treated at the midpoint dose between the not tolerated dose and the last tolerated dose. Zeaxanthin is supplied as 50 milligram capsules and a person's dose will be rounded to the nearest 50 milligrams.
  The dose of pembrolizumab will be administered at a fixed dose of 400 milligrams intravenous every 6 weeks which is an FDA approved dosing schedule to treat cancer patients with pembrolizumab.
  Arms: Zeaxanthin plus Pembrolizumab

SUMMARY:
The purpose of the research is to determine the highest dose of an oral compound called zeaxanthin that can be safely taken each day in patients with advanced cancer, the toxicity profile of zeaxanthin, and the dose of zeaxanthin to use in future cancer clinical trials.

DETAILED DESCRIPTION:
The primary purpose of the study is to determine the safety and optimal dosing of zeaxanthin. Effects on tumor growth will also be looked at but as a secondary endpoint. This study will use a 3+3 design which means that 3 people will receive a certain dose of zeaxanthin and if well tolerated then the next group of people will receive a higher dose. This dose escalation will continue until the highest dose allowed by the study is reached, or a dose is found that is felt not to be safe. If at a given dose one of the three people develops a severe side effect, then three more people will be treated at that dose. If no additional severe side effects develop, then the dose escalation will continue. If two people at a given dose develop severe side effects, that dose will be considered dose limiting and escalation will stop. The doses of zeaxanthin will be based on weight starting with 2 milligrams of zeaxanthin per kilogram of body weight (mg/kg) followed by 4 mg/kg, 6 mg/kg, and finally 8 mg/kg. If a dose level is found to be unsafe, then a new group of patients will be treated at the midpoint dose between the not tolerated dose and the last tolerated dose. Zeaxanthin is supplied as 50 milligram capsules and a person's dose will be rounded to the nearest 50 milligrams.

ELIGIBILITY:
Inclusion Criteria for Dose escalation zeaxanthin monotherapy

1. Stage IV or unresectable stage 3 histologically confirmed solid tumor malignancy refractory to all standard therapies known to provide clinical benefit (unless the therapy is contraindicated or intolerable) in the opinion of the treating investigator for his/her tumor type. Subjects are not required to have received systemic therapies that have response rates under 20% with no associated survival benefit (for example DTIC chemotherapy and high dose Interleukin-2 in melanoma patients).
2. Age ≥ 18 years.
3. Performance status ECOG 0, 1 or 2
4. Adequate organ and marrow function as describe below:

   * Absolute neutrophil count ≥ 1,500/mcL
   * Platelets ≥ 100,000/mcl
   * Total bilirubin < 1.5 x the normal institutional limits excluding patients with confirmed Gilbert's syndrome
   * AST (SGOT)/ALT (SPGT) ≤ 3 x the institutional upper limit of normal (ULN)
   * Creatinine ≤ 1.5 x the institutional upper limit of normal
5. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   Recommended methods of birth control are:
   1. The consistent use of an approved hormonal contraception (birth control pill/patches, rings), An intrauterine device (IUD), Contraceptive injection (Depo-Provera), Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam), Sexual abstinence (no sexual intercourse) or Sterilization.
   2. Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy

   A Female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets at least one of the following criteria:
   1. Has not undergone a hysterectomy or bilateral oophorectomy
   2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
6. Ability to understand and the willingness to sign a written informed consent.
7. Measurable disease is not required but evaluable disease is required.
8. Life expectancy of at least 3 months

Exclusion Criteria for Dose escalation zeoxanthin monotherapy

1. Patients who have had chemotherapy or radiotherapy within 21 days prior to initiating study treatment or those who have not recovered to grade 1 or less from adverse events due to agents administered more than 21 days earlier excluding alopecia, gd 2 fatigue, gd 2 hearing loss from platinum agent, and endocrinopathies on stable replacement therapy.

   (Patients may not be receiving any other investigational agents or concomitant chemotherapy or radiation therapy. Hormonal therapy is not exclusionary.)
2. Patients with active brain metastases requiring palliation with steroids and not stable for at least 4 weeks post radiation therapy or surgery.
3. Leptomeningeal carcinomatosis
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to zeaxanthin.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients with another primary malignancy not in remission for at least 3 years. Exceptions include nonmelanoma skin cancer, curatively treated localized prostate cancer with normal prostate specific antigen, low risk prostate cancer followed expectantly, stage I colorectal cancer resected, resected stage 1 breast cancer cervical carcinoma in situ on biopsy, melanoma in situ resected, or squamous intraepithelial lesion on PAP smear.
7. Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants. Women of child bearing potential must have a negative serum or urine pregnancy test prior to the first dose of study treatment
8. Inability to swallow pills.

Inclusion Criteria for dose escalation zeoxanthin plus pembrolizumab

1. Stage IV or unresectable stage 3 histologically confirmed solid tumor malignancy for which pembrolizumab is FDA approved and progressed on prior PD-1 or PD-L1 therapy and if indicated for cancer type refractory to all standard therapies known to provide clinical benefit (unless the therapy is contraindicated or intolerable) in the opinion of the treating investigator for his/her tumor type. Subjects are not required to have received systemic therapies that have response rates under 20% with no associated survival benefit (for example DTIC chemotherapy and high dose Interleukin-2 in melanoma patients).
2. Patients must have had symptomatic or radiographic progression during or following treatment with a PD-1 or PD-L1 inhibitor. This is defined as imaging obtained subsequent to initiation of PD-1 or PD-L1 inhibitor demonstrating a new lesion that is consistent with metastasis or growth of a preexisting metastasis which the treating physician felt reflected tumor progression and therefore discontinued the immunotherapy. . Symptomatic progression refers to development of worsening bone pain related to bone metastasis that cannot be accurately measured on imaging and for which the treating physician had discontinued the immunotherapy.
3. Age ≥ 18 years.
4. Performance status ECOG 0, 1or 2.
5. Adequate organ and marrow function as describe below:

   * Absolute neutrophil count ≥ 1,500/mcL
   * Platelets ≥ 100,000/mcl
   * Total bilirubin) ≤ 1.5 x normal institutional limits excluding patients with confirmed Gilbert's syndrome
   * AST (SGOT)/ALT (SPGT) ≤ 3 x institutional upper limit of normal
   * Creatinine ≤ 1.5 x the institutional upper limit of normal
6. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   Recommended methods of birth control are:
   1. The consistent use of an approved hormonal contraception (birth control pill/patches, rings), An intrauterine device (IUD), Contraceptive injection (Depo-Provera), Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam), Sexual abstinence (no sexual intercourse) or Sterilization.
   2. Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy

   A Female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets at least one of the following criteria:
   1. Has not undergone a hysterectomy or bilateral oophorectomy
   2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
7. Ability to understand and the willingness to sign a written informed consent.
8. Measurable disease is not required but evaluable disease is required
9. Life expectancy of at least 3 months

Exclusion Criteria for zeoxanthin plus pembrolizumab

1. Patients who have had immunotherapy, chemotherapy or radiotherapy within 21 days prior to entering the study or those who have not recovered to grade1 or lower from adverse events due to agents administered more than 21 days earlier excluding alopecia, gd 2 fatigue, gd 2 hearing loss from platinum agent, and endocrinopathies on stable replacement therapy.
2. Prior grade 3 or greater immune mediated toxicity related to PD-1 or PD-L1 inhibitor. Prior grade 2 or higher colitis, diarrhea, hepatitis, neurologic, cardiac, immune mediated toxicity related to PD-1 or PD-L1 inhibitor. Exceptions include vitiligo and controlled endocrinopathies.
3. Patients may not be receiving any other investigational agents or concomitant chemotherapy or radiation therapy.
4. Patients taking oral steroids at or greater than the equivalent of 10 milligrams of oral prednisone daily.
5. Inability to swallow pills.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to zeaxanthin.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants. Women of child bearing potential must have a negative serum or urine pregnancy test prior to the first dose of study treatment
9. Patients with active brain metastases requiring palliation with steroids not stable for at least 4 weeks post radiation therapy or surgery
10. Leptomeningeal carcinomatosis
11. Patients with another primary malignancy not in remission for at least 3 years. Exceptions include non-melanoma skin cancer, curatively treated localized prostate cancer with normal prostate specific antigen, low risk prostate cancer followed expectantly, resected stage 1 colon cancer, resected stage 1 breast cancer, cervical carcinoma in situ on biopsy, melanoma in situ resected, or squamous intraepithelial lesion on PAP smear.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Zeaxanthin monotherapy | Up to 20 weeks for each dosing cohort
  Recommended maximum tolerated dose
  Highest dose of zeaxanthin that does not cause dose limiting toxicity in patients with unresectable advanced solid tumors treated with zeaxanthin
Zeaxanthin monotherapy (continued) | Toxicities experienced within 28 days of zeoxanthin initiation
  Rate of Dose Limiting Toxicity (DLT) Based on CTEP Active Version (version 5.0) of the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0) in patients with unresectable advanced solid tumors treated with zeaxanthin
Zeaxanthin plus Pembrolizumab | Up to 20 weeks for each dosing cohort
  Recommended maximum tolerated dose
  Highest dose of zeoxanthin that does not cause dose limiting toxicity in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab
Zeaxanthin plus Pembrolizumab (continued) | Toxicities experienced within 42 days of zeaxanthin plus pembrolizumab initiation
  Rate of Dose Limiting Toxicity (DLT)
  Based on CTEP Active Version (version 5.0) of the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0) in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab

SECONDARY OUTCOMES:
The response rate (ORR) of zeaxanthin in patients with unresectable advanced solid tumors | 36 months
  The ORR by RECIST v1.1 of zeaxanthin in patients with unresectable advanced solid tumors Duration of response: duration from date of initial attainment of CR or PR to date of progression, censoring at death or lost to follow-up Disease Control rate: percent of patients who develop CR, PR, or stable disease as best response as determined by RECIST v1.1 measured at 2 months and 6 months after initiation of study treatment Progression Free Survival: duration of time in months from the initiation of study treatment to date of progression, censoring at death or lost to follow-up.
The response rate of zeaxanthin plus pembrolizumab in patients with unresectable advanced solid tumors | 36 months
  The ORR by RECIST v1.1 of zeaxanthin plus pembrolizumab in patients with unresectable advanced solid tumors
The duration of response (DR) in patients with unresectable advanced solid tumors treated with zeaxanthin | 36 months
  The DR by RECIST v1.1 of zeaxanthin in patients with unresectable advanced solid tumors
The duration of response in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab | 36 months
  The DR by RECIST v1.1 of zeaxanthin plus pembrolizumab in patients with unresectable advanced solid tumors
The disease control rate (DCR) in patients with unresectable advanced solid tumors treated with zeaxanthin | Week 8 and Week 24
  Percentage of patients with complete response, partial response, or stable disease according to RECIST v1.1 measured at 2 months and 6 months after initiation of zeaxanthin treatment
The disease control rate (DCR) in patients with unresectable advanced solid tumors treated with zeaxanthin plus zeaxanthin | Week 8 and Week 24
  Percentage of patients with complete response, partial response, or stable disease according to RECIST v1.1 measured at 2 months and 6 months after initiation of zeaxanthin plus pembrolizumab treatment
The progression free survival (PFS) for zeaxanthin in in patients with unresectable advanced solid tumors | Up to 24 months
  The PFS rate for zeaxanthin in patients with unresectable advanced solid tumors as measured by RECIST v1.1
The progression free survival (PFS) for zeaxanthin plus pembrolizumab in in patients with unresectable advanced solid tumors | Up to 24 months
  The PFS rate for zeaxanthin in patients with unresectable advanced solid tumors as measured by RECIST v1.1
The maximal plasma concentration of zeaxanthin in patients treated with zeoxanthin | Pharmacokinetic (PK) sampling will be performed on Day 1, 2, 8, 15,22, 28, 56, 84
  To evaluate the effect of multiple doses of zeaxanthin on the steady state pharmacokinetics of zeoxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin
The maximal plasma concentration of zeoxanthin in patients treated with zeoxanthin plus pembrolizumab | Pharmacokinetic (PK) sampling will be performed on Day 1, 2, 8, 15,22, 43, 64
  To evaluate the effect of multiple doses of zeoxanthin on the steady state pharmacokinetics of zeoxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab
Area under the curve (AUC) of zeaxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin | Pharmacokinetic (PK) sampling will be performed on Day 1, 2, 8, 15,22, 28, 56, 84
  Pharmacokinetics of zeaxanthin as measured by AUC
Area under the curve (AUC) of zeaxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab | Pharmacokinetic (PK) sampling will be performed on Day 1, 2, 8, 15,22, 28, 56, 84
  Pharmacokinetics of zeaxanthin as measured by AUC

OTHER OUTCOMES:
On treatment biopsy for evidence of increased immune cell infiltration and vascularization to zeaxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin | Up to 36 months
  Measured by changes in immune cell populations and CD31 vascularization between baseline and on treatment tumor biopsy specimens
On treatment biopsy for evidence of increased immune cell infiltration and vascularization to zeoxanthin in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab | Up to 36 months
  Measured by changes in immune cell populations and CD31 vascularization between baseline and on treatment tumor biopsy specimens
On treatment percentage changes in immune cell composition in peripheral blood in patients with unresectable advanced solid tumors treated with zeaxanthin | Up to 36 months
  Measured by changes in the percentage of different immune cell populations between baseline and on treatment blood specimens
On treatment percentage changes in immune cell composition in peripheral blood in in patients with unresectable advanced solid tumors treated with zeaxanthin plus pembrolizumab | Up to 36 months
  Measured by changes in percentage of different immune cell populations between baseline and on treatment blood specimens
Changes in blood transcriptome in patients with unresectable advanced solid tumors treated with zeaxanthin | Up to 36 months
  Measured by changes in PBMC samples obtained at baseline and on treatment with PBMCs subjected to bulk RNA sequencing
Changes in blood transcriptome in patients with unresectable advanced solid tumors treated with zeaxanthin plus zeaxanthin | Up to 36 months
  Measured by changes in PBMC samples obtained at baseline and on treatment with PBMCs subjected to bulk RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Philip Friedlander, MD, Principal Investigator — The Valley Hospital
Locations (1):
- The Valley Hospital-Luckow Pavilion, Paramus, New Jersey, United States